CLINICAL TRIAL: NCT04525222
Title: An mHealth Mood Management Tool to Improve Population-Level Cessation
Brief Title: mHealth Mood Management Tool (Actify) to Improve Population-Level Smoking Cessation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Jaimee Heffner, Associate Professor, Fred Hutchinson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RG1121054; NCI-2020-05454 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10540 (Other: Fred Hutch/University of Washington Cancer Consortium); R34DA050967 (NIH)
Record Dates: First submitted 2020-08-13; First posted 2020-08-25 (Actual); Results first posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Cigarette Smoking-Related Carcinoma
MeSH Terms: interventions — Health Promotion; Educational Status; Smoking Devices

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Any outcome evaluator who has direct contact with participants will be blinded to treatment group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (Actify, text notifications) (Experimental): Participants use Actify app for smoking cessation for 8 weeks. Participants also receive motivational messages and smoking cessation information via text notifications.
  Interventions: Other: Health Promotion and Education; Behavioral: Smoking Cessation Intervention (Actify app); Other: Survey Administration
- Arm II (Current Standard Care, text notifications) (Active Comparator): Participants use app for smoking cessation for 8 weeks. Participants also receive motivational messages and smoking cessation information via text notifications.
  Interventions: Other: Health Promotion and Education; Behavioral: Smoking Cessation Intervention (Current Standard Care app); Other: Survey Administration

INTERVENTIONS:
Other: Health Promotion and Education — Receive motivational messages and smoking cessation information via text notifications
Behavioral: Smoking Cessation Intervention (Actify app) — Use Actify app
  Other Names: Smoking and Tobacco Use Cessation Interventions
  Arms: Arm I (Actify, text notifications)
Behavioral: Smoking Cessation Intervention (Current Standard Care app) — Use (USCPG) Current Standard Care app
  Other Names: Smoking and Tobacco Use Cessation Interventions
  Arms: Arm II (Current Standard Care, text notifications)
Other: Survey Administration — Ancillary studies

SUMMARY:
This phase I trial investigates a new smartphone application (called Actify) for improving population-level smoking cessation and mood management. Actify delivers behavioral activation therapy for depression as part of a smoking cessation intervention and will be compared to another smoking cessation smartphone application that is based on current clinical practice guidelines. Participants will be randomly assigned to receive one of two smartphone applications and accompanying text notifications to help with quitting smoking and improved mood.

DETAILED DESCRIPTION:
OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I: Participants use Actify app for smoking cessation for 8 weeks. Participants also receive motivational messages and smoking cessation information via text notifications.

ARM II: Participants use United States (US) Clinical Practice Guidelines (USCPG) app for smoking cessation for 8 weeks. Participants also receive motivational messages and smoking cessation information via text notifications.

After completion of study, participants are followed up at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Current smoker, averaging at least 5 cigarettes/day for the last 30 days
* Interested in quitting smoking in the next 30 days
* Experience downloading and using one or more apps on their smartphone
* Either screens negative (Patient Health Questionnaire - 9 Item [PHQ-9] score 0-4) for depression or screens positive for mild to moderate current depressive symptoms (PHQ-9 score 5-19)
* Willing and able to complete all study activities
* Comfortable reading and writing in English
* Have a mobile data plan and/or access to WiFi to support the use of the Actify app
* Reside in the US
* Have a smartphone either an iPhone (running iOS version 11 or higher) or an Android phone (running version 5.0 or higher)

Exclusion Criteria:

* Currently receiving behavioral treatment for depression (e.g., psychotherapy)
* Current use of a depression app
* Severe depression (PHQ-9 >= 20)
* Receiving other treatment for smoking cessation
* Previous use of the QuitGuide app
* Current or recent (within the past year) enrollment in a Fred Hutch smoking cessation study
* Employees/family of investigator or study center
* Member of the same household as another participant
* Woman who is pregnant or breastfeeding, or planning to become pregnant
* Currently incarcerated
* Is ineligible per fraud prevention protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2023-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaimee Heffner, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two-hundred forty two participants were eligible and enrolled in the study. The final sample comprised 242 participants who were randomized between May 9, 2022 and September 30, 2022.
Period: Overall Study
Arm/Group | Arm I (Actify, Text Notifications) | Arm II (Current Standard Care, Text Notifications)
Started | 119 | 123
Completed | 100 | 98
Not Completed | 19 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Actify, Text Notifications) | Arm II (Current Standard Care, Text Notifications) | Total
Number analyzed (Participants) | 119 | 123 | 242
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.5 (11) | 52 (9.8) | 50.3 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 84 | 167
  Male | 36 | 39 | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 6 | 13
  Not Hispanic or Latino | 112 | 117 | 229
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 4 | 4
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 21 | 38
  White | 95 | 86 | 181
  More than one race | 2 | 7 | 9
  Unknown or Not Reported | 5 | 5 | 10
Smoking Level (in the past 30 days) - High (20+ CIgs/Day) [Count of Participants; unit: Participants] | 64 | 66 | 130
Smoking Level (in the past 30 days) - Low (<20 Cigs/Day) [Count of Participants; unit: Participants] | 55 | 57 | 112
Mental Health Condition - Anxiety, Depression, Bipolar, Schizophrenia, Alcohol or Drug Abuse [Count of Participants; unit: Participants] | 23 | 34 | 57
No Mental Health Condition [Count of Participants; unit: Participants] | 96 | 89 | 185
Cigarettes per Day in the past 30 days) [Mean (Standard Deviation); unit: cigarettes per day] | 18 (7.7) | 20.2 (13.2) | 19.1 (10.9)

OUTCOME MEASURES:

1. Primary Outcome: Overall Satisfaction With Assigned Treatment on the Treatment Satisfaction Survey
Description: Overall treatment satisfaction is reported on a Likert-type scale, with response choices ranging from "not at all=1" to "very much=5". Higher values are associated with higher level of satisfaction.
Time Frame: At 8 weeks post-randomization
Population: Overall number of participants analyzed include those who opened the app at least once AND answered at least one acceptability question in the 8 week follow-up survey.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I (Actify, Text Notifications) | Arm II (Current Standard Care, Text Notifications)
Number analyzed (Participants) | 90 | 94
units on a scale | 4.1 (1.0) | 3.7 (1.1)
Statistical Analysis 1: Comparison: Arm I (Actify, Text Notifications) vs Arm II (Current Standard Care, Text Notifications); Treatment satisfaction items are reported on a Likert-type scale, with response choices ranging from "not at all" to "very much". We used a linear regression adjusting for Treatment Arm, Sex Assigned at Birth, Baseline Level of Smoking (<20 Cigs/ >=20 Cigs), and Baseline Depression Severity (PHQ-8<5 / PHQ-8>=5) to test for differences between arms."; Test type: Other; p = 0.0088, Regression, Linear; Adjusting for Treatment Arm, Sex Assigned at Birth, Baseline Level of Smoking (<20 Cigs/ >=20 Cigs), Baseline Depression Severity (PHQ-8<5 / PHQ-8>=5); Slope = 0.42, 95% CI 2-sided [0.10 to 0.74]

2. Primary Outcome: Application (App) Utilization
Description: Number of app openings during the 8-week treatment period.
Time Frame: At 8 weeks post-randomization
Population: We used negative binomial regression adjusting for Treatment Arm, Sex Assigned at Birth, Baseline Level of Smoking (<20 Cigs/ >=20 Cigs), and Baseline Depression Severity (PHQ-8<5 / PHQ-8>=5) to compare number of app openings by treatment arm
Measure: Mean (Standard Deviation); unit: app openings
Arm/Group | Arm I (Actify, Text Notifications) | Arm II (Current Standard Care, Text Notifications)
Number analyzed (Participants) | 103 | 110
app openings | 34.3 (33.7) | 34.3 (39.4)
Statistical Analysis 1: Comparison: Arm I (Actify, Text Notifications) vs Arm II (Current Standard Care, Text Notifications); Test type: Other; p = 0.75, Negative Binomial Regression; [statistical method as in outcome 1, analysis 1]; Slope = 2.92, 95% CI 2-sided [-15.22 to 21.07]

3. Secondary Outcome: Biochemically-confirmed 30-day PPA From Smoking
Description: Self-reported 30-day smoking abstinence at 8 weeks, confirmed via expired carbon monoxide (CO<6ppm)
Time Frame: At 8 weeks post-randomization
Measure: Number; unit: participants
Arm/Group | Arm I (Actify, Text Notifications) | Arm II (Current Standard Care, Text Notifications)
Number analyzed (Participants) | 119 | 123
participants
  No Quit | 109 | 115
  Quit | 10 | 8
Statistical Analysis 1: Comparison: Arm I (Actify, Text Notifications) vs Arm II (Current Standard Care, Text Notifications); Test type: Other; p = 0.55, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.5 to 3.48]

4. Secondary Outcome: Self-reported 30-day PPA From Smoking
Description: Self-reported 30-day abstinence on the survey question of "Have you smoked at all, even a puff, in the last 30 days?"
Time Frame: At 6 months post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Actify, Text Notifications) | Arm II (Current Standard Care, Text Notifications)
Number analyzed (Participants) | 119 | 123
Participants
  No Quit | 97 | 108
  Quit | 22 | 15
Statistical Analysis 1: Comparison: Arm I (Actify, Text Notifications) vs Arm II (Current Standard Care, Text Notifications); Test type: Other; p = 0.17, Regression, Logistic; Adjusting for Treatment Arm, Sex Assigned at Birth, Baseline Level of Smoking <20 Cigs/ >=20 Cigs, Baseline Depression Severity PHQ-8<5 / PHQ-8>=5; Odds Ratio (OR) = 1.63, 95% CI 2-sided [0.80 to 3.32]

5. Secondary Outcome: Biochemically-confirmed 30-day PPA From Smoking
Description: Self-reported 30-day smoking abstinence at 6 months, confirmed via expired carbon monoxide (CO<6 ppm)
Time Frame: At 6 months post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Actify, Text Notifications) | Arm II (Current Standard Care, Text Notifications)
Number analyzed (Participants) | 119 | 123
Participants
  No Quit | 104 | 113
  Quit | 15 | 10
Statistical Analysis 1: Comparison: Arm I (Actify, Text Notifications) vs Arm II (Current Standard Care, Text Notifications); Test type: Other; p = 0.25, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.63, 95% CI 2-sided [0.70 to 3.81]

6. Secondary Outcome: Self-reported 7-day PPA From Smoking
Description: Self-reported 7-day abstinence on the survey question of "When was the last time you smoked, or even tried, a cigarette?"
Time Frame: At 8 weeks post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Actify, Text Notifications) | Arm II (Current Standard Care, Text Notifications)
Number analyzed (Participants) | 119 | 123
Participants
  No Quit | 93 | 107
  Quit | 26 | 16
Statistical Analysis 1: Comparison: Arm I (Actify, Text Notifications) vs Arm II (Current Standard Care, Text Notifications); Test type: Other; p = 0.07, Regression, Logistic — Adjusting for Treatment Arm, Sex Assigned at Birth, Baseline Level of Smoking (<20 Cigs/ >=20 Cigs), Baseline Depression Severity (PHQ-8<5 / PHQ-8>=5); [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.88, 95% CI 2-sided [0.94 to 3.72]

7. Secondary Outcome: Biochemically Confirmed 7-day PPA From Smoking
Description: Self-reported 7-day abstinence from smoking, confirmed via expired carbon monoxide (CO < 6ppm)
Time Frame: At 8 weeks post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Actify, Text Notifications) | Arm II (Current Standard Care, Text Notifications)
Number analyzed (Participants) | 119 | 123
Participants
  No Quit | 102 | 115
  Quit | 17 | 8
Statistical Analysis 1: Comparison: Arm I (Actify, Text Notifications) vs Arm II (Current Standard Care, Text Notifications); Test type: Other; p = 0.04, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.42, 95% CI 2-sided [1.00 to 5.85]

8. Secondary Outcome: Self-reported 7-day PPA From Smoking
Description: as for outcome 6
Time Frame: At 6 months post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Actify, Text Notifications) | Arm II (Current Standard Care, Text Notifications)
Number analyzed (Participants) | 119 | 123
Participants
  No Quit | 95 | 105
  Quit | 24 | 18
Statistical Analysis 1: Comparison: Arm I (Actify, Text Notifications) vs Arm II (Current Standard Care, Text Notifications); Test type: Other; p = 0.25, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.47, 95% CI 2-sided [0.75 to 2.89]

9. Secondary Outcome: Biochemically Confirmed 7-day PPA From Smoking
Description: Self-reported 7-day abstinence from smoking, confirmed via expired carbon monoxide (CO < 6ppm)
Time Frame: At 6 months post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Actify, Text Notifications) | Arm II (Current Standard Care, Text Notifications)
Number analyzed (Participants) | 119 | 123
Participants
  No Quit | 103 | 113
  Quit | 16 | 10
Statistical Analysis 1: Comparison: Arm I (Actify, Text Notifications) vs Arm II (Current Standard Care, Text Notifications); Test type: Other; p = 0.17, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.78, 95% CI 2-sided [0.77 to 4.12]

10. Secondary Outcome: Self-reported 30-day PPA From Smoking Cigarettes and Other Non-medicinal Nicotine/Tobacco Products, Including E-cigarettes
Description: Self-reported 30-day abstinence on the survey questions of "Have you smoked at all, even a puff, in the last 30 days?" & "In the last 30 days, how often did you use any kind of e-cigarette or vaping product?" & "In the last 30 days, how often did you use any other tobacco products such as chewing tobacco, snus, hookahs, cigars, cigarillos, tobacco pipes, and kreteks?"
Time Frame: At 8 weeks post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Actify, Text Notifications) | Arm II (Current Standard Care, Text Notifications)
Number analyzed (Participants) | 119 | 123
Participants
  No Quit | 105 | 115
  Quit | 14 | 8
Statistical Analysis 1: Comparison: Arm I (Actify, Text Notifications) vs Arm II (Current Standard Care, Text Notifications); Test type: Other; p = 0.15, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.91, 95% CI 2-sided [0.77 to 4.73]

11. Secondary Outcome: Biochemically Confirmed 30-day PPA From Smoking Cigarettes and Other Non-medicinal Nicotine/Tobacco Products, Including E-cigarettes
Description: Self-reported abstinence from cigarettes and other non-medicinal nicotine/tobacco products, including e-cigarettes, confirmed via at home saliva cotinine test and expired carbon monoxide (CO < 6ppm)
Time Frame: At 8 weeks post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Actify, Text Notifications) | Arm II (Current Standard Care, Text Notifications)
Number analyzed (Participants) | 119 | 123
Participants
  No Quit | 112 | 117
  Quit | 7 | 6
Statistical Analysis 1: Comparison: Arm I (Actify, Text Notifications) vs Arm II (Current Standard Care, Text Notifications); Test type: Other; p = 0.68, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.41 to 3.86]

12. Secondary Outcome: Self-reported 30-day PPA From Smoking Cigarettes and Other Non-medicinal Nicotine/Tobacco Products, Including E-cigarettes
Description: Self-reported 30-day abstinence on survey questions of "Have you smoked at all, even a puff, in the last 30 days?" & "In the last 30 days, how often did you use any kind of e-cigarette or vaping product?" & "In the last 30 days, how often did you use any other tobacco products such as chewing tobacco, snus, hookahs, cigars, cigarillos, tobacco pipes, and kreteks?"
Time Frame: At 6 months post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Actify, Text Notifications) | Arm II (Current Standard Care, Text Notifications)
Number analyzed (Participants) | 119 | 123
Participants
  No Quit | 100 | 110
  Quit | 19 | 13
Statistical Analysis 1: Comparison: Arm I (Actify, Text Notifications) vs Arm II (Current Standard Care, Text Notifications); Test type: Other; p = 0.21, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.63, 95% CI 2-sided [0.75 to 3.46]

13. Secondary Outcome: Biochemically Confirmed 30-day PPA From Smoking Cigarettes and Other Non-medicinal Nicotine/Tobacco Products, Including E-cigarettes
Description: as for outcome 11
Time Frame: At 6 months post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Actify, Text Notifications) | Arm II (Current Standard Care, Text Notifications)
Number analyzed (Participants) | 119 | 123
Participants
  No Quit | 107 | 115
  Quit | 12 | 8
Statistical Analysis 1: Comparison: Arm I (Actify, Text Notifications) vs Arm II (Current Standard Care, Text Notifications); Test type: Other; p = 0.30, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.63, 95% CI 2-sided [0.63 to 4.19]

14. Secondary Outcome: Change in Depressive Symptoms Via Patient Health Questionnaire-8 (PHQ-8)
Description: The Patient Health Questionnaire-8 (PHQ-8) is an assessment of depressive symptoms used to detect symptom changes over time as a result of treatment. The PHQ-8 asks the number of days in the past 2 weeks the respondent had experienced a particular depressive symptom. Possible answers are "not at all" or "several days" or "more than half the days" or "nearly every day," with points (0 to 3) assigned to each category. The scores for each item are summed to produce a total score between 0 and 24 points. A total score of 0 to 4 represents no significant depressive symptoms. A total score of 5 to 9 represents mild depressive symptoms; 10 to 14, moderate; 15 to 19, moderately severe; and 20 to 24, severe.
Time Frame: Baseline to 8 weeks
Population: Follow-up score minus baseline score.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I (Actify, Text Notifications) | Arm II (Current Standard Care, Text Notifications)
Number analyzed (Participants) | 98 | 101
units on a scale | .7 (4.2) | 2.2 (5.2)
Statistical Analysis 1: Comparison: Arm I (Actify, Text Notifications) vs Arm II (Current Standard Care, Text Notifications); Test type: Other; p = .0072, Regression, Linear; [statistical method as in outcome 1, analysis 1]; Slope = -1.68, 95% CI 2-sided [-2.90 to -0.46]

15. Secondary Outcome: Self-reported 30-day Point Prevalence Abstinence (PPA) From Smoking
Description: Self-reported 30-day abstinence on the survey question of "Have you smoked at all, even a puff, in the last 30 days?"
Time Frame: At 8 weeks post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Actify, Text Notifications) | Arm II (Current Standard Care, Text Notifications)
Number analyzed (Participants) | 119 | 123
Participants
  No Quit | 104 | 114
  Quit | 15 | 9
Statistical Analysis 1: Comparison: Arm I (Actify, Text Notifications) vs Arm II (Current Standard Care, Text Notifications); Test type: Other; p = 0.1770, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.829, 95% CI 2-sided [0.770 to 4.344]

16. Secondary Outcome: Change in Behavioral Activation Subscale Score on the Behavioral Activation for Depression Scale (BADS)
Description: The Behavioral Activation for Depression Scale (BADS) is a 25-item scale used to track changes in behaviors hypothesized to underlie depression and specifically targeted for change by behavioral activation. BADS items are rated on a 7-point scale ranging from 0 (not at all) to 6 (completely). The behavioral activation subscale contains 7 items, with a scoring range of 0 to 42. Change scores reflect the value of the BADS behavioral activation subscale score at 8-week follow-up minus the baseline score. Positive change values indicate an increase in behavioral activation (i.e, an improvement), whereas negative scores indicate a decrease in behavioral activation.
Time Frame: Baseline to 8 weeks post-randomization
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm I (Actify, Text Notifications) | Arm II (Current Standard Care, Text Notifications)
Number analyzed (Participants) | 98 | 101
score on a scale | -2.4 (9.6) | .8 (8.9)
Statistical Analysis 1: Comparison: Arm I (Actify, Text Notifications) vs Arm II (Current Standard Care, Text Notifications); Test type: Other; p = 0.0025, Regression, Linear; Adjusting for Treatment Arm, Sex Assigned at Birth, Baseline Level of Smoking (<20 Cigs/ >=20 Cigs), Baseline Depression, Baseline Activation Score; Slope = 3.62, 95% CI 2-sided [1.28 to 5.95]

ADVERSE EVENTS:
Time Frame: 3-months
Description: Volunteered adverse events collected throughout the 3-month follow-up.
Arm/Group | Arm I (Actify, Text Notifications) | Arm II (Current Standard Care, Text Notifications)
All-Cause Mortality (participants affected / at risk) | 0/119 | 0/123
Serious Adverse Events (participants affected / at risk) | 0/119 | 0/123
Other Adverse Events (participants affected / at risk) | 0/119 | 0/123

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-13): https://cdn.clinicaltrials.gov/large-docs/22/NCT04525222/Prot_SAP_001.pdf
  • Informed Consent Form (2022-06-26): https://cdn.clinicaltrials.gov/large-docs/22/NCT04525222/ICF_000.pdf